CLINICAL TRIAL: NCT06597513
Title: A Single-Arm Trial of Hematopoietic Stem Cell Transplantation-Supported Dose-Dense Chemotherapy with Adebrelimab As First-Line Treatment for Extensive-Stage Small-Cell Lung Cancer
Brief Title: Auto-HSCT-Supported Dose-Dense Chemotherapy with Adebrelimab As First-Line Treatment for ES-SCLC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC-24-07
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Auto-HSCT; Adebrelimab; Dose-Dense Chemotherapy; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- auto-HSCT-Supported Dose-Dense Chemotherapy With Adebrelimab (Experimental): Complete two 21-days cycles of standard-dose etoposide 80-100 mg/m² on days 1-3 and carboplatin AUC 5-6 on day 1, followed by G-CSF for stem cell mobilization. Receive dose-dense etoposide 160-200 mg/m² on days 1-3 and carboplatin AUC 10-12 on day 1 followed by autologous stem cell reinfusion for two 21-day cycles. If eligible, participants will receive standaed-dose etoposide and carboplatin plus adebrelimab 1200 mg on day 1 for four cycles. Finally, participants may enter a maintenance phase with adebrelimab1200 mg every 21 days.
  Interventions: Drug: auto-HSCT-Supported Dose-Dense Chemotherapy With Adebrelimab

INTERVENTIONS:
Drug: auto-HSCT-Supported Dose-Dense Chemotherapy With Adebrelimab — Induction:
  Two 21-day cycles of standard-dose etoposide 80-100 mg/m² on days 1-3 and carboplatin AUC 5-6 on day 1.
  Those without disease progression will advance to consolidation treatment.
  Consolidation:
  Stem cell mobilization with G-CSF will be start when white blood cell count is at its nadir post-chemotherapy.
  After recovery, peripheral blood stem cells will be collected via apheresis, evaluated, and cryopreserved if adequate.
  Dose-dense etoposide 160-200 mg/m² on days 1-3 and carboplatin AUC 10-12 on day 1 for two 21-day cycles.
  Within 48-72 hours after the first cycle, autologous peripheral blood stem cells will be reinfused with G-CSF.
  Further consolidation will depend on hematopoietic recovery with standard-dose EC plus adebrelimab 1200 mg on day 1 for four 21-day cycles.
  Maintenance:
  Adebrelimab 1200 mg every 21 days will be given until disease progression, intolerable toxicity, death, patient withdrawal, or investigator decision.
  Other Names: auto-HSCT, Dose-Dense Chemotherapy, Adebrelimab

SUMMARY:
The goal of this clinical trial is to learn if hematopoietic stem cell transplantation-supported dose-dense chemotherepy with adebrelimb works to treat extensive-stage small-cell lung cancer in adults. It will also assess the safety of this treatment approach.

The main questions it aims to answer are:

Does hematopoietic stem cell transplantation-supported dose-dense chemotherepy with adebrelimb improve the median progression free survival and 12-months overall survival rates? What medical problems do participants experience whild undergoing this treatment?

Participants will:

Complete two 21-days cycles of standard-dose etoposide and carboplatin, followed by G-CSF for stem cell mobilization.

Receive dose-dense chemotherapy followed by autologous stem cell reinfusion for two 21-day cycles.

If eligible, participants will receive etoposide and carboplatin plus adebrelimab for four cycles.

Finally, participants may enter a maintenance phase with adebrelimab.

Throughout the trial, participants will:

Visit the clinic every 21 days for check-ups and tests. Imaging examination every 6 weeks. Followed up by telephone every 2 months

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed small cell lung cancer (SCLC) staged as extensive-stage (ES-SCLC) according to the Veterans Administration Lung Study Group (VALG) classification.
2. ES-SCLC dose not received prior systemic treatment.
3. History of localized-stage SCLC with prior radiotherapy and chemotherapy, with the requirement for definitive treatment, and a minimum of 6 months interval from the last treatment to diagnosis of ES-SCLC.
4. CT or MRI scan ≤28 days prior to the first dose of study medication, with at least one target lesion that has not been irradiated (RECIST v1.1 criteria).
5. Male or female patients aged ≥18 and ≤70 years.
6. ECOG Performance Status of 0 or 1.
7. Life expectancy ≥12 weeks.
8. Adequate organ system function (excluding use of any blood components or growth factors during screening).
9. Male or female participants must agree to use appropriate contraception (e.g., intrauterine device, contraceptive pills, or condoms) from the start of the study treatment until 6 months after the last study treatment; women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
10. Subjects voluntarily participate in this study and sign the informed consent form (ICF).

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC and NSCLC.
2. Prior treatment with any T-cell co-stimulatory or immune checkpoint inhibitors, including but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, or other T-cell targeted agents.
3. Prior treatment with vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor (VEGFR) inhibitors.
4. Symptomatic brain metastases, leptomeningeal disease, or spinal cord compression. For treated brain metastases, the following criteria must be met: no progression on MRI ≥4 weeks post-treatment, completion of treatment ≥28 days before the first dose of study drug, and no need for systemic corticosteroids (>10 mg/day prednisone or equivalent) ≤14 days before the first dose.
5. Hematologic disorders including, but not limited to, lymphoma, acute or chronic leukemia, multiple myeloma, aplastic anemia, or myelodysplastic syndromes.
6. Symptomatic third-space fluid accumulation, such as uncontrolled pericardial effusion, pleural effusion, or ascites despite drainage or other treatments.
7. Active, known, or suspected autoimmune diseases. Exceptions include vitiligo, type 1 diabetes, autoimmune thyroiditis with only hormone replacement therapy, or conditions unlikely to relapse without external stimuli.
8. Use of systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressants ≤14 days before the first dose of study drug. Inhaled or topical corticosteroids and adrenal replacement therapy are allowed if no active autoimmune disease.
9. Receipt of or planned vaccination with live vaccines ≤4 weeks before the first dose of study drug.
10. Interstitial lung disease, drug-induced pneumonitis, radiation pneumonitis requiring corticosteroids, active pneumonia, or severe pulmonary dysfunction.
11. Active tuberculosis or history of active tuberculosis ≤48 weeks before screening, regardless of treatment status.
12. Toxicities from prior anticancer treatment other than alopecia and fatigue must have resolved to CTCAE v4.03 ≤ Grade 1 before the first dose. Long-term sequelae such as platinum-based neurotoxicity are allowed if anticipated to be stable.
13. Imaging (CT or MRI) showing tumor invasion of major vessels, hemoptysis symptoms within 3 months before screening, or daily hemoptysis ≥2.5 mL.
14. Minor surgery (including catheter placement) ≤48 hours before the first dose of study drug.
15. Current or recent use of aspirin (>325 mg/day) or other nonsteroidal anti-inflammatory drugs known to inhibit platelet function ≤10 days before the first dose.
16. Current or recent use of full-dose oral or parenteral anticoagulants or thrombolytics ≤10 days before the first dose. Preventive anticoagulation is allowed.
17. Known hereditary bleeding disorders or coagulation dysfunction. Significant bleeding symptoms or clear bleeding tendencies (e.g., gastrointestinal bleeding, bleeding ulcers, baseline stool occult blood ++ or more) within 12 weeks before screening.
18. History of thromboembolic events within 24 weeks before signing the ICF, including stroke (including transient ischemic attack, hemorrhagic stroke, or infarction), deep vein thrombosis, or pulmonary embolism.
19. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg), hypertensive crises, or history of hypertensive encephalopathy.
20. History of gastrointestinal ulcers, perforation, corrosive esophagitis or gastritis, inflammatory bowel disease, diverticulitis, abdominal fistula, tracheoesophageal fistula, or intra-abdominal abscess within 24 weeks before signing the ICF.
21. Uncontrolled cardiac symptoms or diseases, including: (1) NYHA Class ≥II heart failure; (2) unstable angina; (3) myocardial infarction within 24 weeks; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
22. Known allergy to study drug or excipients, or a history of severe allergic reactions to any monoclonal antibody.
23. Other malignancies within 5 years before the first dose, except for adequately treated cervical carcinoma in situ, basal cell carcinoma, squamous cell carcinoma of the skin, locally excised prostate cancer, or ductal carcinoma in situ with minimal risk of metastasis and expected cure.
24. Known psychiatric disorders, alcohol abuse, drug abuse, or substance misuse.
25. Positive HBsAg with HBV DNA levels exceeding normal limits (1000 copies/ml or 500 IU/ml), or positive HCV (HCV RNA or HCV Ab indicating acute or chronic infection); known HIV positive or acquired immunodeficiency syndrome (AIDS).
26. Uncontrolled or symptomatic hypercalcemia.
27. Receipt of any investigational drug or participation in another interventional clinical trial ≤4 weeks before signing the ICF.
28. History of allogeneic bone marrow transplantation or solid organ transplantation.
29. Use of systemic immunosuppressive drugs ≤2 weeks before randomization.
30. History of hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, carboplatin, or etoposide.
31. Any other factors that, in the investigator's judgment, may lead to premature discontinuation of the study, including non-compliance, severe concurrent illness (including psychiatric illness), significant laboratory abnormalities, or factors affecting the safety or data collection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Time Frame: Followed up every 21 days.
  Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0, detailed descriptions of the events, the onset timing, severity grade, therapeutic interventions undertaken, and the potential correlation with the investigational medication.

SECONDARY OUTCOMES:
Median Progression Free Survival (mPFS) | Imaging examination every 6 weeks.
  The time of disease progression or death in 50% of patients according to K-M curve.
12-months OS rate | Followed up by telephone every 2 months
  The percentage of patients survival in the 12th months according to the K-M curve.
24-months OS rate | Followed up by telephone every 2 months
  The percentage of patients survival in the 24th months according to the K-M curve.

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, MD, Study Director — The First Affiliated Hospital of Guang Zhou Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu M, Guan W, Xie X, Li Z, Qiu G, Lin X, Xie Z, Zhang J, Qin Y, Huang Z, Xu X, Zhou C. Phase I Clinical Trial of Autologous Hematopoietic Stem Cell Transplantation-Supported Dose-Intensified Chemotherapy With Adebrelimab as First-Line Treatment for Extensive-Stage Small Cell Lung Cancer. Clin Lung Cancer. 2025 May;26(3):e236-e241. doi: 10.1016/j.cllc.2024.12.013. Epub 2024 Dec 27. PMID 39848827